CLINICAL TRIAL: NCT05584631
Title: The Influence of Body Composition on Immunoglobulin Disposition After Intravenous and Subcutaneous Administration
Brief Title: IVIG vs SCIG in CIDP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Luigi Brunetti, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro2019001038
Record Dates: First submitted 2022-10-10; First posted 2022-10-18 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: CIDP; Immunoglobulin Deficiency; Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: immunoglobulin; pharmacokinetics; obesity
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Agammaglobulinemia; Obesity | interventions — Immunoglobulins, Intravenous; Hizentra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous immune globulin G (Experimental): Subjects will receive there current intravenous immune globulin dose.
  Interventions: Drug: Intravenous immune globulin G
- Subcutaneous immune globulin G (Experimental): The dosage will be converted from the subject's current intravenous immune globulin G dosage 1:1 (gm per gm).
  Interventions: Drug: Subcutaneous immune globulin G

INTERVENTIONS:
Drug: Intravenous immune globulin G — Intravenous immune globulin G dosed based on the subjects's current dose received for the treatment of CIDP.
  Other Names: Privigen, IVIG
  Arms: Intravenous immune globulin G
Drug: Subcutaneous immune globulin G — Subcutaneous immune globulin G converted from the subject's current IVIG dose 1:1.
  Other Names: Hizentra, SCIG
  Arms: Subcutaneous immune globulin G

SUMMARY:
Current dosing practices for immunoglobulin G (IgG) may be inadequate in extreme body weight. The current study will evaluate the influence of body composition on intravenous and subcutaneous administration of immunoglobulin G in patients.

DETAILED DESCRIPTION:
Current dosing practices for immunoglobulin G (IgG) may be inadequate in extreme body weight. Total (TBW), ideal (IBW), and adjusted (AdjBW) body weight-based dosing strategies are suggested, but these recommendations are based on expert opinion rather than high quality evidence. The adoption of a specific strategy is highly variable depending on the clinician and/or institutional setting. Recently, payors have also adopted strategies to reduce IgG therapy costs of by capping doses. These recommendations are often based on the presumption that IgG distribution is limited to the vascular space. While this assertion is logical, it does not account for changes adipose tissue may confer on target sites, nor does it account for the potential for adipose tissue to function serve as a metabolic sink or a source of inflammatory mediators. The later would be especially important in patients receiving SCIG. Several observational studies have evaluated IgG dosing in obese patients and have been the source of support for dosing strategies. Many of these studies were not representative of specific populations, contained a wide variety of patients with different IgG indications, and had inadequate serum sampling. More recently, the phase III randomized controlled PATH trial did not find a correlation with serum IgG concentrations and clinical endpoints. However, it is important to note that the study was not designed to evaluate pharmacokinetic and pharmacodynamic endpoints. There is also considerable interpatient variation in response; therefore, identification of patient characteristics that predict response or IgG change from baseline will be a useful tool to improve patient responses. Our study will evaluate the influence of body composition and other patient characteristics may have on IgG exposure when given intravenously or subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with a current diagnosis of CIDP (based on European Federation of Neurological sciences / Peripheral Nerve Society CIDP diagnostic criteria).
* 1:1 conversion of IVIG to SCIG (weekly dose conversion) must fall within 0.2-to-0.4 mg/kg dose for SCIG.

Exclusion Criteria:

* Patients receiving IVIG for indications other than CIDP will be excluded.
* Patients with liver impairment (elevations in liver enzymes of greater than 3 times the upper limit of normal) or reduced renal function (CrCl < 50 mL/min) will be excluded
* Active malignancies
* Diabetes
* Myasthenia gravis
* Immunodeficiency
* Autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-11 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of drug half-life | Through study completion, an average of 4 weeks
  Calculation of drug half-life based on data obtained from serum samples
Assessment of immune globulin G serum concentration after intravenous immune globulin G administration | Just before drug administration, immediately after drug administration, approximately days 7 and 14 post drug administration
  Serum IgG concentration (including subtype) will be measured using a human IgG ELISA kit
Assessment of immune globulin G serum concentration after subcutaneous immune globulin G administration | Just before drug administration, immediately after drug administration, approximately days 2, 4 and 7 post drug administration
  Serum IgG concentration (including subtype) will be measured using a human IgG ELISA kit

SECONDARY OUTCOMES:
Assessment of grip strength | Baseline and just before administration of next immune globulin dose.
  Grip strength will be measured using the handheld Martin Vigorimeter just before each dose of IgG is administered during the study period. Subjects will be asked to squeeze the dynamometer as hard as possible with each of his or her hands in a standing position.
Assessment of muscle function | Baseline and just before administration of next immune globulin dose.
  The Medical Research Council (MRC) system for testing and grading of muscle function aims to provide a standardized and objective way to assess muscle function. It was originally introduced in 1943 and has a long history of use in neurology, rehabilitation and general medicine examinations. Assessments of muscles are done bilaterally, meaning that for each muscle tested, the same muscle on the opposite side of the body is also tested. The MRC sum score is finally calculated by adding the score of each individually assessed muscle. The MRC score ranges from 0 - 30 with 0 as the worst outcome.
Assessment of patient disability | Baseline and just before administration of next immune globulin dose.
  The Rasch Overall Disability scale (I-RODS) and the Inflammatory Neuropathy Cause and Treatment Sensory (INCAT) sum score disability scale will be completed before the infusion of IgG. The I-RODS score can range from 0 to 48 with 0 representing the greatest disability. The INCAT score ranges from 0 - 10 with 10 representing worse outcome.
Assessment of fatigue | Baseline and just before administration of next immune globulin dose.
  Fatigue is a common patient concern in CIDP and the Rasch-built fatigue severity scale (R-FSS) will be completed before the infusion of IgG. The R-FSS ranges from 9 to 63 with 63 being the worst score

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Brunetti, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, The State University of New Jersey Clinical Research Center, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No